CLINICAL TRIAL: NCT04909775
Title: A Prospective, Single Center Clinical Study to Examine Cisplatin-based Chemotherapy Combined With Tislelizumab as Bladder Sparing Treatment for Patients With Muscle Invasive Bladder Cancer
Brief Title: Chemotherapy Combined With Tislelizumab as Bladder Sparing Option for Patients With Muscle Invasive Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJBS-001
Record Dates: First submitted 2021-05-17; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Muscle-Invasive Bladder Carcinoma
Keywords: Bladder sparing treatment; muscle invasive bladder cancer; Tislelizumab; immunotherapy
MeSH Terms: interventions — tislelizumab; spartalizumab; Cisplatin; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Cisplatin-based chemotherapy combined with tislelizumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Patients will receive 4 cycles of Tislelizumab (200mg per cycle) in combination with cisplatin-based chemotherapy before cystectomy discussion. The patients reach clinical complete remission will receive tislelizumab maintenance therapy for a year or 13 cycles.
  Interventions: Drug: Tislelizumab; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Tislelizumab — 200 mg per cycle, IV on day 1 of 3-week
  Other Names: anti-PD-1 monoclonal antibody
Drug: Cisplatin — 70mg/m2 IV on Day 1 of 3-week, for 4 cycles. Dose fractionation is permissible.
  Other Names: cis-platinum
Drug: Gemcitabine — 1000mg/m2, Day 1 and Day 8 of 3-week, for 4 cycles
  Other Names: Gemcitabine Hydrochloride

SUMMARY:
This study is designed prospectively to investigate the safety, efficacy and feasibility of cisplatin-based chemotherapy combined with tislelizumab as bladder sparing treatment for patients with muscle invasive bladder cancer (MIBC) which are eligible for cisplatin. The patients that achieved clinical remission after 4 cycles of cisplatin/gemcitabine and tislelizumab, will receive tislelizumab maintenance therapy for a year or 13 cycles. Tislelizumab, an anti-programmed death protein-1 (PD-1) monoclonal antibody, was engineered to minimize binding to FcγR on macrophages to abrogate antibody-dependent phagocytosis, a mechanism of T-cell clearance and potential resistance to anti-PD-1 therapy. The safety, tolerability, and efficacy of tislelizumab in patients with PD-L1 positive urothelial carcinoma who progressed during/following platinum-containing therapy was proved in a phase 2 trial (CTR20170071).

This trial investigates the efficacy of cisplatin-based chemotherapy combined with Tislelizumab to induce clinical complete remission of muscle invasive bladder cancer and the feasibility to provide bladder sparing treatment for these patients.

DETAILED DESCRIPTION:
The patients that meet the Inclusion and Exclusion Criteria will treat with 4 cycles of cisplatin-based chemotherapy combined with Tislelizumab (200mg per cycle) prior to cystectomy discussion. The patients that show clinical benefit will receive tislelizumab for bladder sparing. Forty patients will be enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤75 years old on day of signing informed consent
* Signing informed consent
* Patients with histologically confirmed muscle-invasive bladder cancer (cT2-T4, N0, M0) and with strong intent to bladder sparing(Patients with mixed histology, predominantly transitional cells, could be enrolled. )
* Patients must be willing to provide a TURBT specimen during screening and prior to enrollment if adequate specimen (FFPE tissue block or 15 unstained slides) from initial TURBT documenting muscle-invasive urothelial bladder cancer is not available.
* ECOG performance status of 0 or 1
* Adequate organ and marrow function for cisplatin treatment
* No received prior therapy with systemic chemotherapy or immunotherapy

Exclusion Criteria:

* Received prior therapies targeting PD-1, PD-L1, PD-L2, CTLA4, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Any approved anticancer therapy within 28 days before enrollment
* Active leptomeningeal disease or uncontrolled, untreated brain metastasis
* Participants with uncontrolled hypercalcemia
* Participants with active autoimmune diseases or history of autoimmune diseases that may relapse
* History of interstitial lung disease, noninfectious pneumonitis, or uncontrolled diseases
* A known history of HIV infection
* Prior allogeneic stem cell transplantation or organ transplantation
* History of severe hypersensitivity reactions to other monoclonal antibodies
* History of allergic reactions to cisplatin, carboplatin, or other platinum-containing compounds

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Clinical complete remission rate (cCR) | Up to 24 months
  The clinical complete remission rate (cCR) was defined as the proportion of patients with clinically confirmed cT0 or cTa(AJCC Cancer Staging Manual,8th ed. 2017 edition ).The cT0 or cTa was assessed by cystoscopy examination at 12 weeks after the initiation of combination therapy. Two-sided Clopper-Pearson 95% confidence intervals were constructed to evaluate the accuracy of cCR.

SECONDARY OUTCOMES:
Duration of cCR | Up to 24 months
  Duration of cCR was defined as the delay between date of reaching cCR and tumour relapse or progression.The status of cCR was evaluated by cystoscopy examination every 3 months after the combination therapy. Stratified Cox proportional hazards models will be used to estimate hazard ratios in all eligible patients.
Bladder-intact event-free survival (BI-EFS) | Up to 24 months
  Bladder-intact event-free survival (BI-EFS) was defined as the time from initiation of combination therapy to the date of occurrence of any following event ：
  1. Recurrence of muscle-invasive bladder cancer based on follow-up cystoscopic evaluation
  2. Lymph node metastases based on CT/MR/PET-CT
  3. Distant metastases based on CT/MR/PET-CT
  4. Bladder cancer-related death
  5. Cystectomy due to any reason
  BI-EFS will be estimated with Kaplan-Meier estimators and corresponding 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Danfeng Xu, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No